CLINICAL TRIAL: NCT03076801
Title: Does Choral Singing Help imprOve Stress in Patients With Ischemic HeaRt Disease?: A Pilot Randomized Controlled Trial
Brief Title: Does Choral Singing Help imprOve Stress in Patients With Ischemic HeaRt Disease?
Acronym: CHOIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Paul MacDonald, Dr. Paul MacDonald, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1019989
Record Dates: First submitted 2017-02-24; First posted 2017-03-10 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Ischemic Heart Disease; Coronary Heart Disease; Myocardial Infarction
Keywords: Choral Singing; Music; Quality of Life; Psychosocial Stress; Cardiac Rehabilitation
MeSH Terms: conditions — Myocardial Ischemia; Coronary Disease; Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator will be blind to participant allocation during chart review at 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choral Singing Intervention (Experimental): In addition to usual medical care, participants in the intervention group will participate in choral singing.
  Interventions: Behavioral: Choral Singing
- Control (No Intervention): The control group will receive usual medical care only. If control group participants join an external singing group during the study period they will not be excluded, but this data will be collected and considered.

INTERVENTIONS:
Behavioral: Choral Singing — In addition to usual medical care, participants in the intervention group will participate in weekly 60-90 minute singing sessions led by professional musicians over a 12-week period. Sessions will begin with a 5-minute physical warm-up of gentle stretching and a 5-minute vocal warm-up. Music will be selected from a variety of genres and eras. Attendance will be taken weekly.
  Arms: Choral Singing Intervention

SUMMARY:
This pilot randomized control trial will examine the role of choral singing on psychosocial stress and cardiovascular outcomes in patients with ischemic heart disease (IHD). The hypothesis is that choral singing will improve psychosocial stress in comparison to the control group and this may have an impact on rates of hospitalization, death, myocardial infarction and stroke in these patients.

DETAILED DESCRIPTION:
Objectives:

The purpose of this pilot study is to examine the impact of choral singing on psychosocial stress and major cardiovascular events in patients with IHD in comparison to usual medical care.

Recruitment and Randomization:

Participants will be recruited from community cardiac rehabilitation programs with recruitment presentations, phone calls and mailed invitations. Interested participants will complete baseline questionnaires and provide consent. They will be randomly allocated to either the intervention or control group. Stratification by past or present experience in organized singing (as a binary variable, yes or no) will be used.

Baseline Assessment:

All participants will undergo a baseline assessment, comprised of biophysical characteristics and medical history; level of physical activity self reported by International Physical Activity Questionnaire (IPAQ) long form; assessment of music appreciation and current participation in group singing; and three questionnaires measuring psychosocial stress: the Perceived Stress Scale (PSS), Hospital Anxiety and Depression Scale (HADS) and the Standard Form - 36 (SF - 36).

Intervention:

Participants in the intervention group will participate in weekly 60-90 minute singing sessions led by professional musicians over a 12-week period. Sessions will begin with a 5-minute physical warm-up of gentle stretching and a 5-minute vocal warm-up. Music will be selected from a variety of genres and eras. Attendance will be taken weekly.

Control:

The control group will receive usual medical care. If control group participants join a singing group during the study period they will not be excluded, but this data will be collected and considered.

Analysis:

Data analysis will be done blind with respect to participant allocation. Analysis will include and account for attendance or adherence to consider dose response. Only participants who have attended at least 50% of group singing sessions will be included. A sub-group comparison between those who have attended 50-74% of sessions and those who have attended ≥75% will be done to determine if there is a dose-response effect to the weekly singing sessions. Participants who join another singing group during or after the intervention period will not be excluded, but this will be taken into account. The concept of music "responders" and "non-responders" will be considered based on the initial screening question "How important is music in your day-to-day life?".

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a history of myocardial infarction or acute coronary syndrome and have undergone cardiac rehabilitation. All levels of musical ability and past experience will be included.

Exclusion Criteria:

* Participants unable to respond to English questionnaires will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Psychosocial Stress | Baseline, 3 months and 6 months
  Change in a composite measure of stress from baseline to 3 months and 6 months is the Primary Outcome Measure. This composite measure of stress is comprised of of the Perceived Stress Scale (PSS), Hospital Anxiety and Depression Scale (HADS) and the Standard Form - 36 (SF - 36). Individual scores for the three scales will be determined for each participant at baseline, 3 and 6 months. These scores will be converted to the same scale and averaged with each component weighted equally to determine the composite stress score for each participant.

SECONDARY OUTCOMES:
Rate of hospitalization. | 12 months
  Rates of hospitalization over 12 months will be determined by chart review.
Rates of death. | 12 months
  Rates of death over 12 months will be determined by chart review.
Rates of myocardial infarction . | 12 months
  Rates of myocardial infarction over 12 months will be determined by chart review.
Rates of stroke. | 12 months
  Rates of stroke over 12 months will be determined by chart review.
Intervention adherence | 3 months
  Weekly attendance will be taken for participants in the intervention arm.

OTHER OUTCOMES:
Qualitative Feedback | 3 months
  As a tertiary outcome, informal, qualitative feedback about the music intervention from intervention participants and the musicians running the sessions will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Paul MacDonald, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Heart and Lung Wellness Centre, Sydney, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No